CLINICAL TRIAL: NCT02291744
Title: A Randomized Phase Ⅱ Study of XELOX Chemotherapy With or Without Surgery of Primary Lesion for Colon Cancer Patients With Unresectable Metastatic Lesions
Brief Title: A Phase Ⅱ Study of XELOX Chemotherapy With or Without Surgery of Primary Lesion for Colon Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Weijian Guo, professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: guoweijian-2014-XELOX
Record Dates: First submitted 2014-11-04; First posted 2014-11-14 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Metastatic Colon Cancer
Keywords: TFS (time to failure of strategy)
MeSH Terms: conditions — Colonic Neoplasms | interventions — XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- XELOX plus surgery (Experimental): Eight cycles of XELOX chemotherapy plus surgery:Oxaliplatin 130mg/m2 ivgtt d1 and capecitabine 1000mg/m2,bid,po,d1-d14,every three weeks for a cycle. After 4 cycles, the patients are randomized to surgery group. Then the rest four cycles are administrated.
  Interventions: Procedure: resection of primary lesion; Drug: XELOX
- XELOX (Active Comparator): Eight cycles of XELOX chemotherapy: Oxaliplatin 130mg/m2 ivgtt d1 and capecitabine 1000mg/m2,bid,po,d1-d14,every three weeks for a cycle
  Interventions: Drug: XELOX

INTERVENTIONS:
Procedure: resection of primary lesion — Oxaliplatin 130mg/m2 ivgtt d1 and capecitabine 1000mg/m2,bid,po,d1-d14,every three weeks for a cycle, and resection of primary lesion with metastatic colon cancer
  Arms: XELOX plus surgery
Drug: XELOX — Oxaliplatin 130mg/m2 ivgtt d1 and capecitabine 1000mg/m2,bid,po,d1-d14,every three weeks for a cycle,

SUMMARY:
The primary endpoint is to evaluate the TFS (time to failure of strategy).

DETAILED DESCRIPTION:
The primary endpoint is to evaluate the time to failure of strategy, that is the second progression time after induction therapy by the use of XELOX regimen, comparing XELOX regimen chemotherapy combined with or without surgical resection of the primary lesion from the time of randomization to maintenance therapy and reapplication of induction therapy, or time to the use of second line strategy (if no reapplication of induction therapy) or time to no further treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 18~75 ears old
2. Pathological diagnosis of colon cancer adenocarcinoma
3. No systemic chemotherapy for metastatic tumors
4. ECOG (Eastern Cooperative Oncology Group) 0-1 and expected survival period for 6 months or more
5. At least one measurable objective tumor lesions
6. ANC≥1.5*109/L；PLT≥90*109/L；HB≥90g/L；TBI≤1.5(UNL); ALT、AST≤2.5ULN；Cr≤1.0(ULN) screening within 7 days
7. Primary and metastatic tumors exist at the same time, and distant metastases are not resectable
8. Patients with voluntary participation, and sign the informed consent

Exclusion Criteria:

1. Operation intervention required for perforation, bleeding and obstruction of intestinal cavity
2. With uncontrollable large pleural or peritoneal effusion
3. Alcohol or drug addictions
4. Malignant tumour of the past five years with other organizations to source, but the full treatment of cervical carcinoma in situ and except skin basal cell carcinoma and squamous cell carcinomas
5. With brain metastasis
6. Multiple primary colorectal carcinoma
7. Pregnancy or breast-feeding women
8. There is an important organ failure or other serious diseases, including coronary artery disease, symptomatic cardiovascular disease or myocardial infarction within 12 months; serious neurological or psychiatric history; severe infection; actively disseminated vascula blood coagulation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
TFS time of failure of strategy (the second progression time after induction therapy, or time to the use of second line strategy (if no reapplication of induction therapy) or time to no further treatment) | the second progression time after induction therapy, or time to the use of second line strategy (if no reapplication of induction therapy) or time to no further treatment. The average time is three years.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Huang M, Yang Y, Li Q, Wang C, Liang L, Zhu X, Zhang W, Chen Z, Huang D, Li W, Zhang X, Zhao X, Qiu L, Geng Q, Yu N, Du W, Sun S, Sheng X, Li X, Guo W. Induction Chemotherapy Followed by Primary Tumor Resection Did Not Bring Survival Benefits in Colon Cancer Patients With Asymptomatic Primary Lesion and Synchronous Unresectable Metastases. Front Oncol. 2022 Jan 31;12:747124. doi: 10.3389/fonc.2022.747124. eCollection 2022. PMID 35174078